CLINICAL TRIAL: NCT03787563
Title: Herbal Tea for a Control of Blood Sugar in Subjects With Early Type 2 Diabetes: A Pilot Randomized Placebo Controlled Crossover Study
Brief Title: Herbal Tea in the Treatment of Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Composite Interceptive Med Science (Industry)
Collaborators: Composite Interceptive Med-Science Laboratories Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CIMED - 001- 2018
Record Dates: First submitted 2018-12-23; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Herbal Tea; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Teas, Herbal

STUDY DESIGN:
Intervention Model Description: all the subjects will receive sequence of different study treatments.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Herbal tea (Active Comparator): One tea bag infusion three times a day each before breakfast, lunch and dinner.
  Interventions: Drug: Herbal Tea
- Placebo Tea (Placebo Comparator): Similar looking tea bag infusion three times a day each before breakfast, lunch and dinner.
  Interventions: Drug: Placebo Tea

INTERVENTIONS:
Drug: Herbal Tea — All participants will be given the intervention in an infusion tea bag. Participant will be instructed to take one tea bag three times a day at before breakfast, lunch and dinner meals. At the time of randomization both active and placebo infusion bag will be provided.There will be one day of washout period after 2 days on treatment.
  Arms: Active Herbal tea
Drug: Placebo Tea — Similar looking inert placebo tea.
  Arms: Placebo Tea

SUMMARY:
Diabetes mellitus is a chronic disease caused by inherited and/or acquired deficiency in production of insulin by the pancreas, or by the ineffectiveness of the insulin produced. It has become a major healthcare problem in India. High-quality, low-cost solutions adapted to the local context are critical to addressing the current crisis in the management of diabetes. Herbal tea consists of tulsi, guava and stevia, which has glucose lowering properties.The aim of this trial is to study the effect of a herbal tea in the glycemic response in the early type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Adults aged over 18 years and having a diagnosis of diabetes and meeting one of the following criteria

1. Fasting Plasma Glucose ≥126 mg/dL, fasting defined as no caloric intake for at least 8 hours, AND
2. 2-h Post load Glucose ≥140 mg/dL during an OGTT. AND
3. Glycosylated haemoglobin (A1C) ≥ 6.5 %.

Exclusion Criteria:

Any one of the following

1. Patients on Insulin therapy.
2. Patients on oral hypoglycemic agents other than metformin
3. Any history suggestive of micro vascular or macro vascular disease - coronary artery disease, stroke, peripheral artery disease or diabetes related retinal changes.
4. Women in child bearing age unable to practice any form of contraception
5. Patients with diagnosis of Anaemia (Hemoglobin <11 g/dl in Female and <13 g/dl in Male)
6. Impaired renal function; estimated glomerular function <60mls/min/1.73m2.
7. Known history of any chronic illness taking regular pharmacological agents.
8. Blood pressure fluctuations exceeding 20 mmHg on 2 subsequent clinic visits or known history of hypotension or bradycardia in last 6 months or taking 3 or more antihypertensive medications regularly in the last 6 weeks
9. Known history of autonomic dysfunction like diabetic autonomic neural imbalance or neuropathy
10. Participating in another clinical trial with an active intervention or drug or device with last dose taken within 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Fasting Plasma Glucose (FPG) | 2 days and 5 days
  Change from baseline in Fasting plasma glucose
Oral Glucose Tolerance Test (OGTT) | 2 days and 5 days
  Change from baseline in OGTT
Number of Subject with adverse events | 2 days and 5 days
  Adverse events is defined as any untoward medical occurrence that may not necessarily have a causal relationship with the treatment, but resulted in a dose reduction or discontinuation of treatment.

SECONDARY OUTCOMES:
Flash Glucose Measurements | 2 days and 5 days
  Change from baseline in mean amplitude glycemic excursions measured by flash glucose monitoring sensor

CONTACTS AND LOCATIONS:
Overall Officials: HD Ramachandra Prabhu, MBBS, MD, Principal Investigator — Health India Hospital
Locations (1):
- Health India Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided